CLINICAL TRIAL: NCT01946477
Title: A Phase 2, Multicenter, Multi-cohort, Open-label Study of Pomalidomide in Combination With Low-dose Dexamethasone or Pomalidomide in Combination With Low-dose Dexamethasone and Daratumumab in Subjects With Relapsed or Refractory Multiple Myeloma Following Lenalidomide Based Therapy in the First or Second Line Setting.
Brief Title: Pomalidomide in Combination With Low-dose Dexamethasone or Pomalidomide in Combination With Low-dose Dexamethasone and Daratumumab in Subjects With Relapsed or Refractory Multiple Myeloma Following Lenalidomide-based Therapy in the First or Second Line Setting
Acronym: POM MM 014
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-014
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma, MM, cancer, oncology, hematology, plasma, neoplasm, plasmacytoma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Plasmacytoma | interventions — pomalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomalidomide + dexamethasone (Experimental): Each subject enrolled in the study will take oral pomalidomide (4 mg) once daily on Days 1-21 and dexamethasone 40 mg/day (< 75 years old) or 20 mg/day (>75 years old) on Days 1, 8, 15 and 22 of a 28-day cycle.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- Pomalidomide + Dexamethasone + Daratumumab (Experimental): Each subject enrolled in the study will take oral pomalidomide (4 mg) once daily on Days 1-21 and dexamethasone 40 mg/day (< 75 years old) or 20 mg/ day (>75 years old) on Days 1, 8, 15 and 22 of a 28-day cycle and daratumumab administered intravenously (IV) at a starting dose of 16 mg/kg at following schedule:
  * Days 1, 8, 15, and 22 of a 28-day cycle for Cycle 1 and Cycle 2
  * Days 1 and 15 for Cycle 3 through Cycle 6
  * Day 1 for Cycle 7 and each cycle thereafter until disease progression
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Pomalidomide
  Other Names: CC-4047
Drug: Dexamethasone
  Other Names: dex
Drug: Daratumumab
  Arms: Pomalidomide + Dexamethasone + Daratumumab

SUMMARY:
This trial will evaluate the efficacy and safety of combination of pomalidomide (POM) and low-dose dexamethasone (LD-Dex) (Cohort A) or the combination of pomalidomide (POM) , daratumumab (DARA) and low-dose dexamethasone (LD-Dex) (Cohort B) in subjects with relapsed or refractory multiple myeloma who have received a first or second line treatment of lenalidomide-based therapy.

This trial will test the hypothesis for Cohort A that the proportion of patients will have an Overall Response Rate (ORR) of > 30 % to reveal that Pomalidomide is efficacious in pretreated patients who are refractory to lenalidomide.

This trial will test the hypothesis for Cohort B that the proportion of patients will have an Overall Response Rate (ORR) of > 70 % to reveal that POM+DARA+LD-Dex is efficacious in pretreated patients who are refractory to lenalidomide.

This trial will test the hypothesis for Cohort C that the proportion of patients will have an Overall Response Rate (ORR) of >60% to reveal that POM+DARA+LD-Dex is efficacious in pretreated patients who are refractory to lenalidomide. This treatment will be in only Japanese patients.

DETAILED DESCRIPTION:
A phase 2, multicenter, multi-cohort, open-label study of pomalidomide in combination with low-dose dexamethasone or pomalidomide in combination with low-dose dexamethasone and daratumumab in subjects with relapsed or refractory multiple myeloma following lenalidomide based therapy in the first or second line setting.

This trial will assess, Overall Response Rate (ORR), Overall Survival (OS), Progression-Free Survival (PFS), Duration of Response (DoR), Time to Response (TTR), Time to Progression(TTP) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  1. Adults (age ≥ 18 years at the time of signing the ICD) with documented diagnosis of MM and measurable disease (serum M-protein ≥ 0.5 g/dL or urine M-protein ≥ 200 mg/24 hours).
  2. Subjects enrolling in Cohort A (POM+LD-dex) must have received 2 prior treatment lines of anti-myeloma therapy. Subjects enrolling in Cohort B and Cohort C (POM+DARA+LD-dex) must have received 1 or 2 prior treatment lines of anti-myeloma therapy.
  3. All subjects must have received prior treatment with LEN or a LEN-containing regimen for at least 2 consecutive cycles as the most recent treatment regimen.
  4. All subjects must have documented disease progression during or after their last antimyeloma therapy.
  5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
  6. Subjects must understand and voluntarily sign an ICD prior to any study related assessments/procedures being conducted.
  7. Subjects must be able to adhere to the study visit schedule and other protocol requirements.
  8. All subjects must provide an adequate bone marrow sample at screening that definitively evaluates the presence or absence of myelodysplastic changes.
  9. Females with child-bearing potential (FCBP†) must agree to use 2 reliable forms of contraception* simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including during dose interruptions), and for at least 28 days after study treatment discontinuation and must agree to regular pregnancy testing during this timeframe. For subjects enrolled in Cohort B and Cohort C, pregnancy prevention and testing will continue until 3 months after last dose of daratumumab.
  10. Females must agree to abstain from breastfeeding during study participation and 28 days after study drug discontinuation. Female subjects enrolled in Cohort B and Cohort C must agree to abstain from breastfeeding and donating eggs during study participation and until 3 months after last dose of daratumumab.
  11. Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 28 days following discontinuation from this study, even if he has undergone a successful vasectomy. Male subjects enrolled in Cohort B and Cohort C must agree to use a latex condom during any sexual contact with FCBP while participating in the study and until 3 months after last dose of daratumumab.
  12. Males must also agree to refrain from donating semen or sperm during the treatment phase and for 28 days after discontinuation from this study treatment. Male subjects enrolled in Cohort B and Cohort C must also agree to refrain from donating semen or sperm during the treatment phase and until 3 months after last dose of daratumumab.
  13. All subjects must agree to refrain from donating blood while on study therapy and for 28 days after discontinuation from this study treatment.
  14. All subjects must agree not to share medication.

      Exclusion Criteria:

      The presence of any of the following will exclude a subject from study enrollment:

  <!-- -->

  1. Any of the following laboratory abnormalities:

     • Absolute neutrophil count < 1,000/μL

     • Platelet count < 75,000/μL for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 30,000/μL for subjects in whom ≥ 50% of bone marrow nucleated cells are plasma cells.

     • Severe renal impairment (Creatinine Clearance [CrCl] < 30 mL/min) requiring dialysis.
     * Corrected serum calcium > 11.5 mg/dL (> 2.8 mmol/L)
     * Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior red blood cell transfusion or recombinant human erythropoietin use is permitted)
     * Serum SGOT/AST or SGPT/ALT > 3.0 x the upper limit of normal (ULN)
     * Serum total bilirubin > 2.0 mg/dL (34.2 μmol/L); or > 3.0 x ULN for subjects with hereditary benign hyperbilirubinemia
  2. Prior history of malignancies, other than MM, unless the subject has been free of the disease for more than 5 years. Allowed exceptions include the following:

     •Basal or squamous cell carcinoma of the skin

     •Carcinoma in situ of the cervix or breast

     • Incidental histological finding of prostate cancer (TNM [tumor, nodes, metastasis] stage of T1a or T1b)
  3. Previous therapy with pomalidomide or daratumumab
  4. Hypersensitivity to thalidomide, LEN, or dex (this includes ≥ Grade 3 rash during prior thalidomide or LEN therapy)
  5. Subjects who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant less than 12 months prior to initiation of study treatment and who have not discontinued immunosuppressive treatment for at least 4 weeks prior to initiation of study treatment and are currently dependent on such treatment.
  6. Subjects with any one of the following:

     • Congestive heart failure (NY Heart Association Class III or IV)
     * Myocardial infarction within 12 months prior to starting study treatment
     * Unstable or poorly controlled angina pectoris, including Prinzmetal's variant angina pectoris
  7. Subjects who received any of the following within 14 days of initiation of study treatment:

     • Major surgery (kyphoplasty is not considered major surgery)

     • Use of any anti-myeloma drug therapy
  8. Use of any investigational agents including for the treatment of multiple myeloma within 28 days or 5 half-lives (whichever is longer) of treatment, unless approved by the sponsor.
  9. Incidence of gastrointestinal disease that may significantly alter the oral absorption of Pomalidomide.
  10. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment
  11. Any serious medical condition, laboratory abnormality, or psychiatric illness, that would preclude participation in the study, or interfere with interpretation of the study results
  12. Pregnant or breastfeeding females
  13. Known human immunodeficiency virus (HIV) positivity; active infectious hepatitis A, B, or C; or chronic hepatitis B or C

      All subjects will be tested for hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (antiHBs), and hepatitis B core antibody (antiHBc). Subjects with the following serological testing are considered not eligible:
      * HBsAg positive
      * HBsAg negative, anti-HBs positive and/or anti-HBc positive and detectable viral DNA

      Note:
      * Subjects who are HBsAg negative, anti-HBs positive, and/or anti-HBc positive, viral DNA negative are eligible. For these subjects, DNA monitoring and prophylactic medication for HBV reactivation are recommended per local practice.
      * Subjects who are seropositive because of hepatitis B virus vaccination are eligible (anti-HBs positive, anti-HBc negative, and HBsAg negative).

      All subjects will be tested for hepatitis C antibody. Subjects are not eligible if known seropositive for hepatitis C virus.

      Note:

      • Subjects who are hepatitis C antibody positive but show no detectable viral RNA for 6 months prior to initiation of study treatment are eligible.
  14. For subjects enrolling in Cohort B and Cohort C - Subject has known allergies, hypersensitivity to mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the Daratumumab IB), or known sensitivity to mammalian-derived products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Approximately 2 years
  The primary endpoint will be the Overall Response Rate (ORR) by modified International Myeloma Working Group (mIMWG) criteria and will be based on the best response prior to the time frame. ORR will consist of the responses of PR or better (Complete Response -CR, Very Good Partial Response-VGPR or Partial Response- PR).

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 7 years
  Overall survival will be calculated as the time from start of treatment until the time of death from any cause. If no death is recorded the subject will be censored at the time the subject was last known to be alive.
Progression-free survival (PFS) | Up to 7 years
  Progression-free survival will be calculated as the time from start of treatment until the time of PD (as determined by the site Investigator based on the mIMWG criteria) or death from any cause on study treatment, whichever comes first. Subjects not experiencing a documented progression will be censored at the time of their last response assessment (or at the time of trial enrollment if no assessment was conducted).
Duration of Response (DoR) | Up to 7 years
  Duration of response, calculated for responders only, is defined as time from the initial documented response (PR or better) to the first confirmed PD or until death from any cause. Subjects without a documented progression will be censored at the time of their last response assessment
Time to Response (TTR) | Up to 2 years
  Time to response, calculated for responders only, is calculated as the time from the start of treatment to the first documented response (PR or better) based on modified International Working Group ( mIMWG) criteria.
Time to progression (TTP) | 6 months after 100% enrollment and 5 years from Last Patient First Visit
  Time to progression will be calculated as the time from start of treatment until PD (as determined by the site Investigator based on the mIMWG criteria) or death from progressive disease. Subjects not experiencing a documented progression will be censored at the time of their last response assessment (or at the time of trial enrollment if no assessment was conducted).
Adverse Events | Up to 7 years
  Number of participants with adverse events including secondary primary malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (49):
- United States (33):
  - Local Institution - 126, Tucson, Arizona
  - Local Institution - 137, Greenbrae, California
  - Local Institution - 109, Los Angeles, California
  - Local Institution - 104, Pleasant Hill, California
  - Local Institution - 108, Whittier, California
  - Local Institution - 138, Denver, Colorado
  - Local Institution - 120, Stamford, Connecticut
  - Local Institution - 145, Jacksonville, Florida
  - Local Institution - 127, Orlando, Florida
  - Local Institution - 133, Pembroke Pines, Florida
  - Local Institution - 136, St. Petersburg, Florida
  - Local Institution - 134, Fairway, Kansas
  - Local Institution - 142, Topeka, Kansas
  - Local Institution - 124, Louisville, Kentucky
  - Local Institution - 103, Westminster, Maryland
  - Local Institution - 146, Gross Pointe, Michigan
  - Local Institution - 102, Kansas City, Missouri
  - Local Institution - 110, St Louis, Missouri
  - Local Institution - 118, East Orange, New Jersey
  - Local Institution - 101, Hackensack, New Jersey
  - Local Institution - 129, Glens Falls, New York
  - Local Institution - 149, The Bronx, New York
  - Local Institution - 130, Durham, North Carolina
  - Local Institution - 123, Cleveland, Ohio
  - Local Institution - 121, Cleveland, Ohio
  - Local Institution - 115, Cleveland, Ohio
  - Local Institution - 122, Mayfield Heights, Ohio
  - Local Institution - 107, Hershey, Pennsylvania
  - Local Institution - 135, Chattanooga, Tennessee
  - Local Institution - 131, Nashville, Tennessee
  - Local Institution - 128, Lubbock, Texas
  - Local Institution - 143, Plano, Texas
  - Local Institution - 106, Spokane, Washington
- Canada (8):
  - Local Institution - 113, Calgary, Alberta
  - Local Institution - 144, Surrey, British Columbia
  - Local Institution - 114, Vancouver, British Columbia
  - Local Institution - 139, Moncton, New Brunswick
  - Local Institution - 140, St. John's, Newfoundland and Labrador
  - Local Institution - 112, Toronto, Ontario
  - Local Institution - 148, Toronto, Ontario
  - Local Institution - 117, Montreal, Quebec
- Japan (7):
  - Local Institution - 205, Fukuoka
  - Local Institution - 208, Kamogawa
  - Local Institution - 204, Kyoto
  - Local Institution - 202, Nagoya
  - Local Institution - 203, Okayama
  - Local Institution - 206, Shibukawa-shi, Gunma-ken
  - Local Institution - 207, Toyohashi
- Local Institution - 119, San Juan, Puerto Rico

REFERENCES:
- [Background] Pelligra CG, Parikh K, Guo S, Chandler C, Mouro J, Abouzaid S, Ailawadhi S. Cost-effectiveness of Pomalidomide, Carfilzomib, and Daratumumab for the Treatment of Patients with Heavily Pretreated Relapsed-refractory Multiple Myeloma in the United States. Clin Ther. 2017 Oct;39(10):1986-2005.e5. doi: 10.1016/j.clinthera.2017.08.010. Epub 2017 Sep 28. PMID 28967482
- [Derived] Bahlis NJ, Siegel DS, Schiller GJ, Samaras C, Sebag M, Berdeja J, Ganguly S, Matous J, Song K, Seet CS, Acosta-Rivera M, Bar M, Quick D, Anz B, Fonseca G, Chung W, Lee K, Mouro J, Agarwal A, Reece D. Pomalidomide, dexamethasone, and daratumumab immediately after lenalidomide-based treatment in patients with multiple myeloma: updated efficacy, safety, and health-related quality of life results from the phase 2 MM-014 trial. Leuk Lymphoma. 2022 Jun;63(6):1407-1417. doi: 10.1080/10428194.2022.2030477. Epub 2022 Feb 8. PMID 35133221
- [Derived] Pierceall WE, Amatangelo MD, Bahlis NJ, Siegel DS, Rahman A, Van Oekelen O, Neri P, Young M, Chung W, Serbina N, Parekh S, Agarwal A, Thakurta A. Immunomodulation in Pomalidomide, Dexamethasone, and Daratumumab-Treated Patients with Relapsed/Refractory Multiple Myeloma. Clin Cancer Res. 2020 Nov 15;26(22):5895-5902. doi: 10.1158/1078-0432.CCR-20-1781. Epub 2020 Sep 14. PMID 32928795
- [Derived] Siegel DS, Schiller GJ, Song KW, Agajanian R, Stockerl-Goldstein K, Kaya H, Sebag M, Samaras C, Malek E, Talamo G, Seet CS, Mouro J, Pierceall WE, Zafar F, Chung W, Srinivasan S, Agarwal A, Bahlis NJ. Pomalidomide plus low-dose dexamethasone in relapsed refractory multiple myeloma after lenalidomide treatment failure. Br J Haematol. 2020 Feb;188(4):501-510. doi: 10.1111/bjh.16213. Epub 2019 Oct 6. PMID 31588567
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com